CLINICAL TRIAL: NCT05963035
Title: Clinical Application of 18F-PFPN PET Imaging in Diagnosis and Staging of Clear Cell Sarcoma of Soft Tissue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0409
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Clear Cell Sarcoma of Soft Tissue
MeSH Terms: conditions — Sarcoma, Clear Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-PFPN PET (Experimental): A positron probe for the targeted melanin
  Interventions: Drug: 18F-PFPN

INTERVENTIONS:
Drug: 18F-PFPN — For patients clinically suspected or confirmed clear cell sarcoma of soft tissue, integrated PET/MR or PET/CT imaging will be performed using targeted melanin-specific imaging agent 18F-PFPN. Meanwhile, multiple parameters will be compared with the general imaging agent 18F-FDG.
  Other Names: 18F-PEG3-FPN

SUMMARY:
This study is a prospective monocentric study aimed to evaluate the diagnosis and staging value of 18F-PFPN PET in clear cell sarcoma of soft tissue. Patients with clinically suspected or confirmed clear cell sarcoma of soft tissue will be recruited and 18F-PFPN PET/MR imaging will be performed. PET/CT imaging will be performed in patients with contraindications to MR. Additionally, to compare the diagnostic efficacy with the traditional imaging agent 18F-FDG, patients will also undergo 18F-FDG PET imaging, and the two imaging intervals will be completed two days apart. The general information, clinical data, 18F-PFPN and 18F-FDG PET/MR or PET/CT imaging results and other imaging data of the patients will be collected. The histopathology of the biopsy or surgical specimen, follow-up and other imaging examinations will be taken as evaluation references. This study plans to set the sample size as 10 cases.

DETAILED DESCRIPTION:
Clear cell sarcoma of soft tissue is a rare malignancy derived from neural crest cells that contain melanin and/or melanin precursors. Melanin is an important target for the diagnosis of clear cell sarcoma of soft tissue. 18F-PFPN, a highly specific melanin-targeting positron probe, has been proven to have excellent pharmacokinetic properties and good biological safety, and can sensitively detect tiny melanin-containing lesions. Therefore, 18F-PFPN PET imaging is expected to be used in diagnosing and staging clear cell sarcoma of soft tissue.

This study was designed as a prospective study to explore the diagnosis and staging value of 18F-PFPN PET in clear cell sarcoma of soft tissue. In this study, patients with clinically suspected or confirmed clear cell sarcoma of soft tissue will be recruited to undergo 18F-PFPN PET/MR imaging. PET/CT imaging will be performed in patients with contraindications to MR. The general information, clinical data, imaging data and histopathology results of patients will be collected. The efficiency of diagnosis and staging of 18F-PFPN was evaluated by comparing the gold standard pathological diagnosis and the general metabolic imaging agent 18F-FDG.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 years or above), regardless of gender;
* Patients with clinically suspected or confirmed clear cell sarcoma of soft tissue (supporting evidence including visual examination, MRI, CT, ultrasound, and histopathological examination, etc.) ;
* Patients who agree to undergo both 18F-PFPN and 18F-FDG PET imaging.

Exclusion Criteria:

* Acute systemic diseases and electrolyte disturbances;
* Patients who plan to get pregnant within six months or are pregnant or breastfeeding;
* The patient or his/her legal representative is unable or unwilling to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 18F-PFPN PET for diagnosis and staging of clear cell sarcoma of soft tissue | 1 years
  18F-PFPN and 18F-FDG PET/MR or PET/CT images will be analyzed by at least 2 physicians experienced in nuclear medicine and radiology. The general information, clinical, histopathological and imaging data of patients will be collected and analyzed to calculate the sensitivity and specificity of 18F-PFPN for diagnosis and staging in clear cell sarcoma of soft tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China

REFERENCES:
- [Derived] Zhang X, Kang F, Zheng H, Gai Y, Wang J, Lan X. Melanin-targeted [18F]-PFPN PET imaging may shed light for clear cell sarcoma. Eur J Nucl Med Mol Imaging. 2023 Dec;51(1):196-201. doi: 10.1007/s00259-023-06439-2. Epub 2023 Sep 16. PMID 37714979